CLINICAL TRIAL: NCT04596215
Title: Benefit of the Oxygen Reserve Index for Control of Success of Preoxygenation in Adults
Acronym: PRIORI
Status: Completed | Type: Observational
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Nina Pirlich, Dr. med., Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: PRIORI 1.0
Record Dates: First submitted 2019-05-31; First posted 2020-10-22 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Preoxygenation
Keywords: Anaesthesia; Preoxygenation; blood gas analysis; Oxygen Reserve Index; Decarboxylation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Valuation of the probability for a correct detection of paO2 < 100 mmHg and paO2 > 200 mmHg using the Oxygen Reserve Index

DETAILED DESCRIPTION:
As mentioned above

ELIGIBILITY:
Inclusion Criteria:

* Indication of an elective surgery with invasive arterial blood pressure measurement in awake patients
* written informed consent

Exclusion Criteria:

* Emergency surgery
* Patients with expected difficult airway and indication for an awake fiberoptic intubation and therefore no need of preoxygenation
* no written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult awake patients for elective surgery with indication for an invasive arterial blood pressure measurement
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Validation of the probability for a correct detection of paO2 < 100 mmHg and paO2 > 200 mmHg using the Oxygen Reserve Index | preoxygenation of 3 minutes
  As mentioned above

SECONDARY OUTCOMES:
Patient characteristics | 48 hours
  age, sex, weight, pre-existing conditions
MAP | preoxygenation of 3 minutes
  mean arterial pressure
NIRS (Near-infrared spectroscopy) | preoxygenation of 3 minutes
  cerebral O2 saturation in %, rSO2C
PI | preoxygenation of 3 minutes
  perfusion index

CONTACTS AND LOCATIONS:
Locations (1):
- Johannes Gutenberg - Universität, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No